CLINICAL TRIAL: NCT04870567
Title: High Dose Rate Brachytherapy vs Stereotactic Ablative Body Therapy in Patients With Early-intermediate Prostate Cancer
Brief Title: HDR Brachytherapy vs SABR in Early-intermediate Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Principal Investigator, Galina Kireeva, Scientific secretary, N.N. Petrov National Medical Research Center of Oncology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2021-03-29; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Biochemical Relapse Free Survival; Complications Rates (Erectile Dysfunction, GI, GU Complications)
Keywords: brachytherapy; stereotactic ablative radiotherapy; survival; complications
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose rate brachytherapy (Active Comparator): After spinal anesthesia steel or plastic needle placement performed under TRUS guidance. Pre- and post-insertion ultrasound based planning is obligatory in all cases. Two fractions of 13Gy are delivered with 2 separate implantations and 2-3 weeks interval. The CTV was defined as the prostate capsule with 1mm (low-risk) - 3 mm (intermediate risk) expansion plus proximal 1/3 of seminal vesicles. The PTV was equal to CTV. The rectum, bladder and urethra are contoured as organs at risk. The dosimetry plan objectives are the following: prostate D90 - above 104% and V100% - above 92%; urethra D10 < 110% , rectum D2cc<75% (below 75Gy EQD2).
  Interventions: Radiation: High dose rate brachytherapy
- Stereotactic ablative radiotherapy (Experimental): Before SBRT three fiducial markers are obligatory inserted into the prostate.Planning MRI on diagnostic table with subsequent fusing with simulation CT is obligatory. CTV to planning target volume (PTV) expansion was 3-5 mm in all direction except posteriorly (in the direction of the rectum) where it is 1-3 mm. Dose must be delivered as 5 fraction of 7.25Gy. V100% for PTV ≥ 95%. Main dose constraints are as follows: D 2cm³ ≤ 36Gy for rectum (below 75Gy EQD2)., V 37.5 Gy <5 cm³ for bladder, V 20 Gy <10 cm³ for femoral heads. Androgen deprivation therapy is not permitted.
  All treatments must be performed on conventional linear accelerators with cone beam CT guidance before each fraction, intrafractional motion monitoring is optional.
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — Patients were randomly assigned (1:1) to conventionally high dose rate brachytherapy or stereotactic body radiotherapy. Randomisation was done Chief researcher blinded to patient data by telephone stratification by risk group (low or intermediate).
  Arms: Stereotactic ablative radiotherapy
Radiation: High dose rate brachytherapy — Patients were randomly assigned (1:1) to conventionally high dose rate brachytherapy or stereotactic body radiotherapy. Randomisation was done Chief researcher blinded to patient data by telephone stratification by risk group (low or intermediate).
  Arms: High dose rate brachytherapy

SUMMARY:
This is single center prospective phase 2 randomized trial aiming to compare biochemical and clinical relapse free survival and toxicity profiles of stereotactic body radiotherapy (SBRT) versus high dose rate brachytherapy (HDRB) for localized low- and intermediate risk prostate cancer patients.

DETAILED DESCRIPTION:
Before SBRT three fiducial markers are obligatory inserted into the prostate. Simulation and every SBRT sessions are performed after bowel preparation (enema) and bladder filling (400ml).Planning MRI on diagnostic table with subsequent fusing with simulation CT is obligatory. The clinical target volume (CTV) include the prostate only (low-risk patients) or prostate and proximal 1/3 of seminal vesicles (intermediate-risk patients). CTV to planning target volume (PTV) expansion was 3-5 mm in all direction except posteriorly (in the direction of the rectum) where it is 1-3 mm. Dose must be delivered as 5 fraction of 7.25Gy. V100% for PTV ≥ 95%. Main dose constraints are as follows: D 2cm³ ≤ 36Gy for rectum (below 75Gy EQD2)., V 37.5 Gy <5 cm³ for bladder, V 20 Gy <10 cm³ for femoral heads. Androgen deprivation therapy is not permitted.

All treatments must be performed on conventional linear accelerators with cone beam CT guidance before each fraction, intrafractional motion monitoring is optional.

After spinal anesthesia steel or plastic needle placement performed under TRUS guidance. Pre- and post-insertion ultrasound based planning is obligatory in all cases. Two fractions of 13Gy are delivered with 2 separate implantations and 2-3 weeks interval. The CTV was defined as the prostate capsule with 1mm (low-risk) - 3 mm (intermediate risk) expansion plus proximal 1/3 of seminal vesicles. The PTV was equal to CTV. The rectum, bladder and urethra are contoured as organs at risk. The dosimetry plan objectives are the following: prostate D90 - above 104% and V100% - above 92%; urethra D10 < 110% , rectum D2cc<75% (below 75Gy EQD2).

Patients are assessed during treatment, 4-12 weeks after the end of the treatment, every 3 months for the first year and then every 6 months till the end of the study. Normal tissue adverse events are reported according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0). International prostate symptoms score (IPSS) and international index of erectile function (IIEF-5) must be assessed on each visit, maximal urinary rate and residual urine volume - annually.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status of 0-2,
* histologically confirmed prostate adenocarcinoma: Gleason score - 6-7 (4+3), clinical stage T1c-T2c, N0, M0
* T and N stage determined by clinical examinations, MRI and/or PET-CT with PSMA
* PSA below 20 ng/ml within the last 30 days
* international prostate index score (IPSS) below 16
* medically fit to spinal anesthesia
* prostate volume below 110 cm³
* maximal urinary rate above 9 ml/sec, residual urine volume below 30ml,
* in the case of previous transurethral resection interval of at least 9 months after procedure.

Exclusion Criteria:

* stage T3-T4,
* PSA > 20 ng/ml,
* clinically detected lymph node or distant metastases,
* previous pelvic irradiation,
* rectal surgery.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer can be detected only in male patients
Enrollment: 350 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of grade 3-5 Adverse Events Assessed by Common Terminology Criteria for Adverse Events CTCAE v5 | 5 years after treatment
  To evaluate frequency of grade 3-5 toxicity in patients treated by high dose rate brachutherapy (arm 1) and stereotactic ablative radiotherapy (arm 2)
Change in the proportion of patients with moderate and severe erectile dysfunction | 3, 6, 12, 18, 24 and every 6 months through 5 years
  Assessed by International Index of Erectile Function (IIEF)

SECONDARY OUTCOMES:
Biochemical relapse free survival | 5 years after treatment
  PSA levels in the blood. Reccurence - nadir + 2 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Sergey Novikov, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided